CLINICAL TRIAL: NCT00499486
Title: Phase II Clinical, Biological and Pharmacological Study of Rapamycin (Rapamune®, Sirolimus) in Patients With Advanced Pancreatic Cancer
Brief Title: Sirolimus in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHOC-J0415, CDR0000549899; P30CA006973 (NIH); JHOC-J0415; JHOC-04-06-16-01
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Sirolimus 5mg. po QD continously (28 days=cycle)
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — Treatment with rapamycin will begin on Day 1 at a single flat dose level of 5 mg/day. Rapamycin will be administered continuously without interruption through all cycles in an outpatient setting. Each cycle will last 28 days.
  Other Names: rapamycin

SUMMARY:
RATIONALE: Sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well sirolimus works in treating patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of patients with previously treated advanced pancreatic cancer surviving at 6 months after treatment with single agent rapamycin.
* To evaluate the relationship between activation of the PI3/Akt/mTOR/S6K signaling pathway in tumor tissues and rapamycin activity in this patient population.
* To characterize toxicity of rapamycin in this patient population.

Secondary

* To determine the response rate, median time to treatment failure, and median survival of patients with previously treated advanced pancreatic cancer who are treated with single agent rapamycin.
* To characterize the pharmacokinetics of rapamycin in this patient population.
* To explore pharmacogenomic variables that affect rapamycin pharmacokinetics and clinical activity in this patient population.
* To determine the pharmacodynamic effects of rapamycin on S6 kinase activation in PBMC, normal skin, and normal oral mucosa obtained from patients treated with the drug and its relationship with rapamycin pharmacokinetics and clinical effects.
* To explore biomarkers in tumor tissues that might be associated with rapamycin clinical effects.

OUTLINE: Patients receive oral sirolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood, normal skin, and tumor tissue collection at baseline and periodically during study for pharmacological, biological, and genotyping studies. Blood samples are analyzed by LC/MS/MS assay to assess rapamycin pharmacokinetics (PKs) during courses 1 and 2 and to determine baseline CYP3A4 activity. Samples are also analyzed by genotyping studies to assess CYP3A4 polymorphisms. Pharmacodynamic activity of rapamycin is assessed in peripheral blood mononuclear cells isolated from PK blood samples using a kinase assay to measure S6K activity. Tumor tissue is collected from pretreatment tumor samples obtained at the time of diagnosis or surgery or by biopsy from patients for whom pre-study tumor specimens are not available. Patients undergo skin biopsies at baseline and on day 1 of course 2 to obtain samples of normal skin. Patients also undergo oral mucosa smears at baseline and weekly during course 1. Tumor tissue, normal skin, and oral mucosa samples are assessed by IHC staining of S6K and p-S6K and by RT-PCR for cyclin D1 and p27.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically proven adenocarcinoma of the pancreas

  * Locally-advanced or advanced disease which has progressed after one prior gemcitabine-containing regimen
* Unidimensionally measurable disease (defined as at least one unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan) OR evaluable disease
* Tumor tissue available for IHC assessment OR willingness to undergo a safe biopsy of tumor tissue

Exclusion criteria:

* Histologic or cytologic diagnosis that is not consistent with adenocarcinoma, including adenosquamous, islet cell, cystadenoma or cystadenocarcinoma, carcinoid, or small or large cell carcinoma or lymphoma
* Adenocarcinoma arising from a site other than the pancreas (e.g., distal common bile duct, ampulla of vater or periampullary duodenum)
* Known brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* WBC > 3,500 cells/mm³
* ANC > 1,500 cells/mm³
* Hemoglobin > 9 g/dL
* Serum creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2 mg/dL
* ALT, AST, and alkaline phosphatase ≤ 5 times upper limit of normal
* Triglycerides and total cholesterol < 2 times upper limit of normal
* Not pregnant or nursing

Exclusion criteria:

* Uncontrolled medical conditions that could potentially increase the risk of toxicities or complications of this therapy, including immunodeficiency and chronic treatment with immunosuppressors
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Active infections
* History of concurrent malignancy or history of a second malignancy within the past 5 years
* Clinically significant cardiovascular disease, including myocardial infarction (within 12 months prior to randomization), unstable angina, grade II or greater peripheral vascular disease, uncontrolled congestive heart failure, or uncontrolled hypertension (i.e., systolic blood pressure (BP) > 170 mm Hg, diastolic BP > 95 mm Hg)

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Any unresolved chronic toxicity greater than CTCAE grade 2 from previous anticancer therapy
* Any previous surgery, excluding minor procedures (e.g., dental work or skin biopsy) within 4 weeks of enrollment
* Participation in an investigational new drug trial within 1 month of starting trial
* Treatment with chemotherapy within 30 days of day 1 treatment
* At least 10 days since prior and no concurrent:

  * Cyclosporine
  * Diltiazem
  * Ketoconazole
  * Rifampin
  * St. Johns wort
  * Grapefruit juice
* Concurrent phenytoin, carbamazepine, barbiturates, or phenobarbital
* No other concurrent investigational or commercial agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garrido-Laguna I, Tan AC, Uson M, Angenendt M, Ma WW, Villaroel MC, Zhao M, Rajeshkumar NV, Jimeno A, Donehower R, Iacobuzio-Donahue C, Barrett M, Rudek MA, Rubio-Viqueira B, Laheru D, Hidalgo M. Integrated preclinical and clinical development of mTOR inhibitors in pancreatic cancer. Br J Cancer. 2010 Aug 24;103(5):649-55. doi: 10.1038/sj.bjc.6605819. Epub 2010 Jul 27. PMID 20664591

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During baseline evaluation (approximately 72 hours prior to treatment with rapamycin), patients will receive a single dose of 3 mg oral midazolam as phenotypic evaluation of CYP3A4 activity.
Groups:
- Sirolimus: Patients with advanced pancreatic adenocarcinoma refractory to gemcitibine received Sirolimus at a single oral flat dose of 5 mg. per day. A treatment cycle was 28 days.
Period: Overall Study
Arm/Group | Sirolimus
Started | 47
Completed | 31
Not Completed | 16
Not completed — Withdrawal by Subject | 16

BASELINE CHARACTERISTICS:
Population: All patients had previously progressed to a gemcitabine-containing regimen, including 22 patients who had received previous chemotherapy for metastatic disease.
Groups:
- Sirolimus: adencarcinoma refractory to gemcitibine
Arm/Group | Sirolimus
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Overall Survival at 6 Months
Time Frame: 6- month survival rate (6mSR)
Measure: Number; unit: % of participants
Groups:
- One Group: Patients with advanced pancreatic adenocarcinoma refractory to gemcitabine
Arm/Group | One Group
Number analyzed (Participants) | 31
% of participants | 26

2. Primary Outcome: Response Rate (Complete, Partial Response and Stable Disease) as Assessed by RECIST
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Response for Stable disease was assessed at 2 months and for complete and partial response at 6 months.
Time Frame: response at 2 and 6 months
Measure: Number; unit: participants
Arm/Group | One Group
Number analyzed (Participants) | 31
participants
  complete and partial response at 6 months | 0
  stable disease at 2 months | 4

3. Primary Outcome: Severity of Adverse Events as Assessed by NCI CTCAE v3.0
Time Frame: 6 months
Measure: Number; unit: percentage of Adverse Events
Arm/Group | One Group
Number analyzed (Participants) | 31
percentage of Adverse Events
  Grade 1 | 67
  Grade 2 | 24
  Grade 3 | 9
  Grade 4 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 7/31
Other Adverse Events (participants affected / at risk) | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=31)
Failure to thrive (General disorders) | 2 (2)
Hyperglycemia (Endocrine disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=31)
elevated Alkaline Phosphatase (Metabolism and nutrition disorders) | 2 (2)
elevated ALT (Metabolism and nutrition disorders) | 4 (7)
Anemia (Blood and lymphatic system disorders) | 9 (11)
Anorexia (Gastrointestinal disorders) | 5 (7)
elevated AST (Metabolism and nutrition disorders) | 5 (8)
Constipation (Gastrointestinal disorders) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
elevated creatinine (Renal and urinary disorders) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 2 (3)
diarrhea (Gastrointestinal disorders) | 4 (4)
Dry mouth (General disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 2 (2)
fatigue (General disorders) | 12 (12)
hyperglycemia (Metabolism and nutrition disorders) | 18 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 12 (13)
lymphopenia (Blood and lymphatic system disorders) | 12 (15)
Mucositis (Gastrointestinal disorders) | 5 (7)
nausea (Gastrointestinal disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 12 (12)
abdominal pain (Gastrointestinal disorders) | 6 (6)
thrombocytopenia (Blood and lymphatic system disorders) | 12 (12)
pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 14 (14)
vomiting (Gastrointestinal disorders) | 3 (3)
hyperchoesterolaemia (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes